CLINICAL TRIAL: NCT06834204
Title: ACCESS-PC: Advancing Care Coordination to Enhance Shared Care for Complex Cancer Survivors in Primary Care.
Brief Title: Advancing Care Coordination Between Cancer and Primary Care Teams for Complex Cancer Survivors
Acronym: ACCESS-PC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Denalee O'Malley, Assistant Professor Rutgers RWJ Medical School Dept Family Medicine and Community Health, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2024000262
Record Dates: First submitted 2025-02-04; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Breast Cancer Early Stage Breast Cancer (Stage 1-3); Bladder Cancer; Prostate Cancer (Adenocarcinoma); Endometrial Cancer; Hypertension; Hyperlipidemia (E.G., Hypercholesterolemia); Diabetes Mellitus
Keywords: primary care; cancer; cardiovascular; shared care; care coordination; implementation; cancer multi-team system; complex cancer survivor
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Adenocarcinoma; Endometrial Neoplasms; Hypertension; Hyperlipidemias; Hypercholesterolemia; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients in this arm will not receive the intervention.
- Primary Care Connect (PC2) (Experimental): Patients enrolled in this arm will be provided print and video educational materials about the importance of shared care to manage existing and prevent exacerbations in chronic disease management. Additionally, their cancer care team will provide a brief protocolized communication to their primary care team that explain how their initial treatment may impact chronic disease management, clarifying the primary care role during acute treatment, and providing contact information for cancer team. Primary care providers of patients enrolled in this arm will receive an outreach packet that includes information provided in print and short video to explain the rationale of the intervention and the materials provided by the cancer care team.
  Interventions: Other: PC2: Primary Care Connect

INTERVENTIONS:
Other: PC2: Primary Care Connect — Primary Care Connect is a health system intervention that includes patient education, electronic medical record optimization, protocolized communication from cancer care team to primary care.
  Arms: Primary Care Connect (PC2)

SUMMARY:
The purpose of this randomized clinical trial is to learn if 'complex' cancer patients who receive care guided by a health system intervention, Primary Care Connect (PC2) have their risks of cardiovascular disease (CVD) managed better than those who receive usual care. This study focuses on "complex" cancer survivors who have higher CVD risk when diagnosed with cancer because they also have had a diagnosis of 1 or more chronic conditions (e.g., hypertension, diabetes, and/or hyperlipidemia) requiring medication management. This study also aims to learn about the ease of implementing the health system intervention from the perspectives of cancer teams, primary care teams, and complex cancer patients.

The main questions the study aims to answer are:

* Do patients enrolled in the PC2 arm remain connected to their primary care teams during active cancer treatment for chronic disease management compared to patients in usual care?
* Do patients enrolled in the PC2 arm have better management of their chronic conditions during active cancer treatment compared to patients in usual care?
* How do the care team and patients experience this change in care delivery related to their work and care experiences?

This study will compare complex cancer survivors who receive care according to the PC2 intervention to usual care to see if PC2 works to improve cardiovascular risk management.

Participants will:

* receive educational materials about the study upon enrollment
* complete on-line or written surveys at 4 times
* Visit the clinic for check ups and test related to the study 4 times

DETAILED DESCRIPTION:
Cancer survivors with cardiovascular disease risk factors (complex cancer survivors) are a growing population and their morbidity and mortality risks are significant. A shared care model (when two or more clinicians of different specialties care for the same patient) is the optimal care delivery model for complex cancer survivors and has been shown to produce optimal comorbidity management when primary care is involved.

Results from our ongoing and recent research studies indicate that survivors managing chronic conditions should not be disconnected from their primary care team. Therefore, feasibility issues must be addressed using stakeholder-informed strategies to enhance the translational potential of shared care that aligns multiple stakeholders (i.e., cancer care team, patients, primary care teams) understandings of this paradigm of care and build team-based care capacities.

This study employs a design-for-dissemination, theory guided perspective, blending implementation science and care delivery conceptual frameworks--Exploration, Planning, Implementation, and Sustainment (EPIS) and Cancer Multi-team System (cMTS)--to understand and address the multi-level factors of implementing shared care in a health system. These perspectives will shape tailoring and implementation of Primary Care Connect (PC2), a health system intervention designed to align complex cancer survivors, healthcare team members, and health system implementation actors' understandings, capacities, and practices to promote the adoption of shared care delivery models for complex cancer survivors.

Using a hybrid type III effectiveness-implementation design this study aims to: (1) engage diverse primary care and health system stakeholders to tailor PC2 to maximize implementation strategies fit to the health system and primary care practice contexts; (2) conduct a randomized controlled trial (n=266 patients) to test the effectiveness of PC2 on primary care connection, chronic disease management, and patient-reported outcomes; and, (3) evaluate PC2 implementation using a mixed methods approach to inform sustainable usage of the intervention. Study results are poised to have a profound impact on the adoption of shared care delivery models throughout the U.S. to optimally mitigate complex cancer survivors CVD risks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with any of the following cancers [Stage I-III]: breast, prostate, urinary bladder, and endometrial in the past 6 months;
* being treated for cancer with curative intent;
* had initial patient visit at the cancer center in the last 3 months;
* are being treated for cancer with curative intent at the Rutgers Cancer Institute of New Jersey
* have ≥1 CVD risk factor (hypertension, hyperlipidemia or type II diabetes) prior to cancer diagnosis that requires medication management;
* currently receiving care from a primary care provider or willing to initiate seeing a new primary care provider upon enrollment;
* Speak English or Spanish

Exclusion Criteria:

* had myocardial infarction or stroke within the previous 1 year; (2) have heart failure with an ejection fraction <30%; (3) have stage IV-V chronic kidney disease (eGFR <30); or do not speak English or Spanish. Patients whose cancer progresses to metastatic disease during the course of the 18-month trial will be allowed to continue to participate unless they voluntarily withdraw

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Connected Care-Continuity with Primary Care Provider | From the time of enrollment to 18-months post enrollment.
  Three primary care visits focused on chronic disease management from time of enrollment to 18-months post-enrollment.

SECONDARY OUTCOMES:
HEDIS quality measure of management hypertension | Baseline, 6-months, 12-months, and 18-months
  blood pressure <140/90mm Hg
HEDIS quality measure of management diabetes | Baseline, 6-months, 12-months, and 18-months
  A1c<8.0%
HEDIS quality measure of management of statin use | Baseline, 6-months, 12-months, and 18-months
  Statin use if patient is diabetic or has a 10-year ASCVD risk >10%. To evaluate statin use, the research team will measure fasting laboratory lipid profile at the time of each study assessment.

OTHER OUTCOMES:
Self-efficacy for Managing Chronic Conditions and Patient Centered Communication | Baseline, 6-months, 12-months, and 18-months
  Self-efficacy for managing chronic conditions: the PROMIS measures will be used to assess and individual's confidence in his/her ability to successfully perform specific tasks or behaviors related to one's health in a variety of situations assessing five domains: daily activities, symptoms, medications and treatments, emotions and social interactions.
  Patient centered communication with both the cancer and primary care teams will be assessed using the validated 7-item scale. We will adapt this scale slightly to use a 6-month recall period given intensity of care during the active cancer and our planned assessment intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Dena O'Malley, PhD, MSW, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers RWJ Medical School, Somerset, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
The cleaned, item-level spreadsheet data for all variables will be shared openly, along with example quantifications and transformations from initial raw data. The rationale for sharing only cleaned data is to foster ease of data reuse.
  The final dataset will include self-reported demographic and behavioral data from participant surveys, interviews, and medical data from lab values and chart abstractions. We will share de-identified individual-participant level (IPD) data. Appropriate measures such as deleting or masking personal identifiers (for quantitative data), and generating quasi-identifiers (e.g., participant names in qualitative interviews) will be used for data de-identification and sharing, and informed consent forms will reflect those plans. All datasets that can be shared will be deposited in Dataverse, an NIH supported data sharing resource and generalist repository, managed by Harvard university.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Shared data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 10 years after the end of the funding period.
Access Criteria: Access/distribution/reuse of the resulting health system implementation actor scientific data (i.e., implementation planning group transcripts, interviews, nurse diaries) will be limited because even after de-identification, individuals, teams and organizations would be inferentially identifiable based on the context. Access to these data will be approved/monitored by the study PIs.
  Survey data and clinical trial data will be de-identified and contextual identifiers will be removed prior to sharing. All sharing will comply with local, state and federal laws and regulations, including HIPAA Privacy and Security Rules. Data will be de-identified before presentations and publications, as well as any datasets shared with qualified researchers who have obtained appropriate IRB approvals.
URL: https://dataverse.harvard.edu/